CLINICAL TRIAL: NCT06886581
Title: Effectiveness of Online Training Course to Improve Evidence-based Leadership Practices: a Cluster Randomised Two-arm Controlled Trial
Brief Title: Online Training Course to Improve Evidence-based Leadership
Acronym: EVILEAD
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Turku (Other)
Collaborators: City of Helsinki (Other); Hospital District of Helsinki and Uusimaa (Other)
Responsible Party: Principal Investigator, Maritta Välimäki, Professor, University of Helsinki
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: Ethics Committee 1/2025; HU 73715712 (Other: University of Helsinki)
Record Dates: First submitted 2025-03-14; First posted 2025-03-20 (Actual); Last update posted 2025-06-13 (Actual); Status verified 2025-06

CONDITIONS: Evidence-Based Practice; Leadership
Keywords: cluster randomised trial; evidence-based; leadership

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Evidence-based leadership training (Experimental): The participants in the experimental group will join a seven months online course aiming to improve the evidence-based leadership competences.
  Interventions: Behavioral: Evidence-based leadership training
- Passive control group (No Intervention): A passive control group

INTERVENTIONS:
Behavioral: Evidence-based leadership training — The structure of the course will follow the steps of the evidence-based approach: (1) each participant will identify their specific unit problem to be solved together with the team and unit leader will work with this problem during the course; (2) organisational data will be collated and analysed to understand the key problem of the unit; (3) scientific literature will be searched for, and critically appraised; (4) the views of stakeholders (patients, family members, etc.) will be considered along with implications; and (5) all sources of information will be collated together and the solution will be implemented into practice; the real situation will be evaluated. Each module includes specific learning material (power points, scientific articles), peer-group discussions, clinical exercises, and self-assessment and self-reflection. The unit leaders will work together their unit members. The course will be run in small group (about 15/agroup) and supported by tutors.
  Arms: Evidence-based leadership training

SUMMARY:
The goal of this cluster clinical trial is to evaluate the effectiveness of online training course, targeted to unit leaders to improve staff's evidence-based skills (individual outcomes), EBP implementation (team-based outcomes), and the quality of care (organisational outcomes). Feasibility and fidelity of the intervention will be assessed as well. The main questions it aims to answer are:

1. Does online training course improve staff's evidence-based practice?
2. Does online training course improve staff's self-esteem and self-efficacy?
3. Does online training course improve leadership for EBP implementation on organisational level?
4. Does online training course improve the quality of patient care?
5. Does online training course reduce staff's absence (sick leaves, intention to leave the ward or hospital)?

Participants will:

* Participants will join in a seven-months online training course in small group or practice as usual.
* Seven course modules, read course material, prepare assignments, join in peer discussions.
* Self-assessment, self-reflection and give course feedback.

DETAILED DESCRIPTION:
This cluster randomisation study will evaluate the effectiveness of online training course, targeted to unit leaders. The intervention will be delivered at the level of the cluster, i.e. professionals within clusters (education of unit leaders). Cluster randomisation study fits our purposes because our intention is to enhance the application of evidence by entire unit teams; the whole groups of collections of individuals in ward units are randomly assigned to receive educational intervention in groups, referred to as clusters.

This cluster trial will be conducted in two Finnish Wellbeing Services counties in southern Finland. The target group of study are unit leaders working in social and health care sector in a managerial position.

The units will be randomised into two groups: evidence-based leadership training (experimental group) or passive control group. The participants in the experimental group will join a seven months online course aiming to improve the evidence-based leadership competences.

All eligible unit leaders who have shown their interest to participate the study will receive an invitation email from the contact person of the study (the Chief Executive Officer). The email will include a link to study information and electronic informed consent in the Research Electronic Data Capture tool (REDCap). After given an electronic informed consent, the REDCap will lead to a baseline survey (background information of the participants of the specific units, baseline data). Unit leaders will be allocated into the study group as their unit.

All staff members who are working in the same unit with the unit leaders will be invited to join the study. First, staff members will receive an invitation email (sent by a Contact person) to explain the purpose of the study and its practical arrangements. If the staff member is willing to join the study, she or he will give an electronic content (REDCap) and respond to electronic surveys - but they do not join online training. After filling electronic forms, each staff members will be allocated into the same study group as their unit.

The outcomes are targeted to evaluate the effectiveness of the evidence-based online course on individual, team, and organisational level. The data will be formed based on characteristics of the unit and its participants, outcome data, course feedback, and feasibility data of the online training course. The primary endpoint with respect to effectiveness of the training course are an improvement in EBP from baseline to follow-up (month 7), measured immediately after the intervention using electronic survey administered to the unit leaders and staff.

The analysis will be carried out on an intent-to-treat (ITT) basis. Assumptions of normality of the residuals will be investigated. The characteristics of the units and respondents (staff members) will be summarized with descriptive statistics for each group. All individuals within the cluster will be included in the trial. In the sample size calculation, a clustering effect was assumed and accounted as the ICC coefficient. For data analysis the mixed effects model or two-level multilevel models that take into account clustering effects will be used. In the model analysis, the variation in the outcomes among clusters will be estimated and tested for its significance. The intra-cluster coefficient (ICC) will be reported. The overall efficacy of the outcomes will be estimated after taking into account the clustering effects. A descriptive summary of the baseline information for both clusters and individuals will be presented first as tables of summary data. Sensitivity analyses will be conducted on units in which participation in online training was low to evaluate whether intervention fidelity has any effect to the results of the primary outcome. Results will be expressed using rate ratios, odds ratios, or least-squares mean differences with corresponding 95% CIs, depending on the type of outcome. The intracluster (or intraclass) correlation coefficient (ICC) will also be calculated.

Covariate analysis will be conducted to control for potential confounding factors in statistical modelling. Participants' age, gender, and the number of returned task (by each participant in intervention group) will be included in the analysis.

ELIGIBILITY:
Inclusion Criteria:

* have shown their willingness to join the study,
* unit leaders have an official managerial position at the study organisation,
* unit have a leaders with a professional licence to work in health or social care sector,
* unit leaders represent any gender,
* are able to speak, read and write in Finnish, and
* have given informed consent to join the study.

Exclusion Criteria:

* Those staff members who are off duty during the recruitment period (family leave, long-term sick leave, study leave, or any other reason).

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2025-06-05 (Actual); Primary Completion 2026-07-01 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
The Evidence-based Practice Questionnaire (EBPQ) | From enrollment to the end of training at 7 months.
  The Evidence-based Practice Questionnaire (EBPQ) assess the implementation of evidence-based practice (24 items, score 1-7, three sub-scales: 1) the knowledge/skills (14 items, score 1-7, 1=Poor-7=Best, the range 14-98, a higher score represents greater knowledge in EBP); 2) the attitudes (4 items, score 1-7, the range 4-28; a higher score represents more a positive attitude toward EBP; 3) an evidence-based practice (6 items, score 1-7, 1=Never, 7=Frequently, range 6-42); the higher score is better.

SECONDARY OUTCOMES:
Self-Esteem Scale (RSE) | From enrollment to the end of training at 7 months.
  Self-Esteem Scale (RSE) evaluate individual self-esteem with a 10-item unidimensional scale by focusing on both positive and negative feelings about the self (4-point Likert scale, 1=strongly agree - 4=strongly disagree). The sum score varies between 10 to 40: the higher score is better and represent higher self-esteem.
The General Self-Efficacy Scale (GSE) | From enrollment to the end of training at 7 months.
  The General Self-Efficacy Scale (GSE) assess optimistic self-beliefs for coping with a variety of difficult demands in life with 10 items (a 4-point Likert scale, 1 = not at all true, 4 = exactly true). Summed score ranges 10 - 40: the higher score indicates better coping abilities.
The Implementation Leadership Scale (ILS) - Staff version | From enrollment to the end of training at 7 months.
  The Implementation Leadership Scale (ILS)- Staff version, is 12-item questionnaire measuring leadership for EBP implementation. It consists of four subscales: (1) proactive leadership, (2) knowledgeable leadership, (3) supportive leadership, and (4) perseverant leadership. It is scored from 0 (not at all) to 4 (to a very great extent); the higher total score represents stronger implementation of EBP.
The Implementation Leadership Scale (ILS) - Supervisor version | From enrollment to the end of training at 7 months.
  The Implementation Leadership Scale (ILS)- Supervisor versions is 12-item questionnaire measuring leadership for EBP implementation. It consists of four subscales: (1) proactive leadership, (2) knowledgeable leadership, (3) supportive leadership, and (4) perseverant leadership. It is scored from 0 (not at all) to 4 (to a very great extent); the higher total score represents stronger implementation of EBP.
The quality of care: Number of Patient Deaths (Register Data) | From enrollment to the end of training at 7 months.
  Number of patient deaths during a seven-month follow-up period reported in hospital registers; lower numbers overall are better.
The quality of care: Number of Treatment Complaints (Register Data) | From enrollment to the end of training at 7 months.
  Number of patient/family members' treatment complaints during a seven-month follow-up period reported in hospital registers; lower numbers overall are better.
The quality of care: Number of Medication Errors (Register Data) | From enrollment to the end of training at 7 months.
  A number of medication errors during a seven-month follow-up period reported in hospital registers; lower numbers overall are better.
Work absence: Number of Staff Absence Days (Register Data) | From enrollment to the end of training at 7 months.
  Number of staff's absence days during a seven-month follow-up period reported in hospital registers (e.g. sick leave); lower numbers overall are better.
Intention to leave the ward - survey | From enrollment to the end of training at 7 months.
  During the last six months, how often a respondent has planned to leave the ward using a five-point scale (0 = never; 1 = now and then; 2 = quite often; 3 = very often; 4 = all the time): lower score is better.
Intention to leave hospital - survey | From enrollment to the end of training at 7 months.
  During the last six months, how often a respondent has planned to leave the hospital using a five-point scale (0 = never; 1 = now and then; 2 = quite often; 3 = very often; 4 = all the time): lower score is better.
Intention to leave profession - survey | From enrollment to the end of training at 7 months.
  During the last six months, how often a respondent has planned to leave the profession using a five-point scale (0 = never; 1 = now and then; 2 = quite often; 3 = very often; 4 = all the time): lower score is better.

OTHER OUTCOMES:
Course feedback - survey | After the course, at month 7.
  Course feedback survey for the participants in experimental group (8 items): 1) "This course was appealing to me"; 2) "I felt happy when I participated in the course"; 3) "Participation in the course required too much effort from me"; 4) "It was worth participating in this course"; 5) "I found this course valuable"; 6) "I was able to meet the requirements of the course"; 7) "This course fits well with my personal values"; and 8) "I would recommend the course to others". Participants will consider the propositions with five possible answers (1 = completely disagree; 2 = disagree; 3 = neither agree nor disagree; 4 = agree; 5 = completely agree): higher total score is better.
Feasibility and fidelity: number of total loggs in each module (f) | After the course, at month 7.
  Number of total loggs in each course module (f) will be calculated; higher total score is better.
Feasibility and fidelity: number of participants who logged in each module (n) | After the course, at month 7.
  Number of the participants will be calculated in Moodle platform who logged in each module (n); higher number of participants is better.
Feasibility and fidelity: adherence to the course (f) | After the course, at month 7.
  Number of returned course tasks (f) out of all possible tasks will be calculated; higher number of returned course tasks is better.
Feasibility and fidelity: adherence to the course tasks (n) | After the course, at month 7.
  Number of participants who returned course tasks by each module (n) will be calculated; higher number of participants who returned course tasks is better.
Feasibility and fidelity: drop-out from intervention | After the course, at month 7.
  Number of participants who leave the intervention early will be calculated (n).
Feasibility and fidelity: drop-out rate of study | After the course, at month 7.
  Number of participants who leave the study early (n) will be calculated (no follow-up data; lower number of participants is better.

CONTACTS AND LOCATIONS:
Overall Officials: Maritta A Välimäki, PhD, Professor, Principal Investigator — University of Helsinki
Locations (1):
- City of Helsinki, Helsinki, South Finland, Finland

IPD SHARING:
Plan to Share IPD: No
Research data will include personal information of the participants. Thereore, entire research data cannot be make publicly available as it is. Meta-data of the study will be published.

REFERENCES:
- [Background] Hu S, Chen W, Satamo M, Loyttyniemi E, Yang M, Liu G, Chen J, Tang Y, Varpula J, Li X, Valimaki M. Online training to improve evidence-based leadership competencies among nurse leaders in China: a feasibility randomised controlled trial. BMJ Open. 2024 Nov 7;14(11):e088386. doi: 10.1136/bmjopen-2024-088386. PMID 39510773
- [Background] Valimaki MA, Kirsi H, Yang M, Lantta T, Varpula J, Liu G, Tang Y, Chen W, Hu S, Chen J, Loyttyniemi E, Li X. Online training to improve evidence-based leadership competencies among nurse leaders in Finland and China: study protocols for two randomised feasibility trials. BMJ Open. 2023 Aug 14;13(8):e067306. doi: 10.1136/bmjopen-2022-067306. PMID 37580090
- [Derived] Valimaki M, Satamo M, Yang M. Effectiveness of an online training course to improve evidence-based leadership practices among unit leaders: study protocol for a cluster randomised two-arm controlled trial (EVILEAD). Trials. 2025 Nov 14;26(1):508. doi: 10.1186/s13063-025-09207-9. PMID 41239490
- See also: Description of the Department — https://www.helsinki.fi/fi/koulutusohjelmat/terveydenhuollon-kehittamisen-maisteriohjelma/opiskelu